CLINICAL TRIAL: NCT04980274
Title: Impact of Admission SOFA Score and 48-hour Delta SOFA on Clinical Outcomes in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, MD; PhD, Hospital Sao Domingos
Other Study IDs: 51
Record Dates: First submitted 2021-07-18; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Critically Ill Patients
Keywords: SOFA SCORE; Delta SOFA; Critically ill patients; Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with SOFA score < 2 on admission
  Interventions: Other: Intervention focused on identified organ dysfunction(s)
- Group 2: Patients with SOFA score equal to or > 2 on admission and who improved after 48 hours of treatment
  Interventions: Other: Intervention focused on identified organ dysfunction(s)
- Group 3: Patients with SOFA score equal to or > 2 on admission and who did not improve after 48 hours of treatment
  Interventions: Other: Intervention focused on identified organ dysfunction(s)

INTERVENTIONS:
Other: Intervention focused on identified organ dysfunction(s) — Intervention focused on identified organ dysfunction(s)

SUMMARY:
Organ dysfunctions are associated with high morbidity and mortality. The SOFA (Sequential Organ Failure Assessment) score developed by Vincent et al. sequentially assesses the presence and severity of dysfunctions in six organ systems: respiratory, cardiovascular, coagulation, hepatic, neurological and renal. Although the SOFA score was created to quantify organ dysfunctions, the obvious relationship between organ dysfunctions and mortality has been widely documented. Dynamic measurements of the SOFA score assess response to treatment and can be used to search for perpetuating sources of severity and reassess the treatment plan.

The primary objective of this study will be to assess the impact of an admission SOFA score equal to or greater than 2 and subsequent interventions on outcomes related to the 48-hour delta SOFA on ICU and hospital mortality, length of stay in the ICU, duration of mechanical ventilation, time of vasoactive drug use.

Patients will be divided into three groups: those who did not trigger the SOFA trigger on admission to the ICU (Group 1), those who triggered the SOFA trigger and improved on the third day (Group 2) and, finally, those who triggered the SOFA trigger and worsened on the third day (Group 3).

ELIGIBILITY:
Inclusion Criteria:

* Included all patients over 18 years old admitted to the ICU during the study period

Exclusion Criteria:

* Excluded were patients who remained in the ICU for a period of less than 48 hours and pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The SOFA score of all patients admitted to the ICU and with inclusion criteria was calculated and whenever the score was equal to or > 2, the attending physician was notified, the dysfunction(s) that resulted in the score was informed and the physician was asked to inform through the therapeutic plan the interventions it would adopt to improve the result after 48 hours
Sampling Method: Probability Sample
Enrollment: 1410 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement in SOFA score after 48 hours of ICU stay | 48 hours
  Interventions designed to reverse or improve the organ dysfunction that motivated a SOFA score equal to or > 2

SECONDARY OUTCOMES:
28 day mortality | 28 days
  Interventions designed to reverse or improve the organ dysfunction that motivated a SOFA
Length of time without mechanical ventilation | 28 days
  Interventions designed to reverse or improve the organ dysfunction that motivated a SOFA
Length of time without vasopressor | 28 days
  Interventions designed to reverse or improve the organ dysfunction that motivated a SOFA

CONTACTS AND LOCATIONS:
Overall Officials: JOSE AZEVEDO, MD, PhD, Study Director — HOSPITAL SAO DOMINGOS SAO LUIS, BRAZIL
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Azevedo JR, Torres OJ, Beraldi RA, Ribas CA, Malafaia O. Prognostic evaluation of severe sepsis and septic shock: procalcitonin clearance vs Delta Sequential Organ Failure Assessment. J Crit Care. 2015 Feb;30(1):219.e9-12. doi: 10.1016/j.jcrc.2014.08.018. Epub 2014 Sep 10. PMID 25241933
- [Result] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Result] Moreno R, Vincent JL, Matos R, Mendonca A, Cantraine F, Thijs L, Takala J, Sprung C, Antonelli M, Bruining H, Willatts S. The use of maximum SOFA score to quantify organ dysfunction/failure in intensive care. Results of a prospective, multicentre study. Working Group on Sepsis related Problems of the ESICM. Intensive Care Med. 1999 Jul;25(7):686-96. doi: 10.1007/s001340050931. PMID 10470572
- [Result] Jones AE, Trzeciak S, Kline JA. The Sequential Organ Failure Assessment score for predicting outcome in patients with severe sepsis and evidence of hypoperfusion at the time of emergency department presentation. Crit Care Med. 2009 May;37(5):1649-54. doi: 10.1097/CCM.0b013e31819def97. PMID 19325482
- [Result] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Result] Raith EP, Udy AA, Bailey M, McGloughlin S, MacIsaac C, Bellomo R, Pilcher DV; Australian and New Zealand Intensive Care Society (ANZICS) Centre for Outcomes and Resource Evaluation (CORE). Prognostic Accuracy of the SOFA Score, SIRS Criteria, and qSOFA Score for In-Hospital Mortality Among Adults With Suspected Infection Admitted to the Intensive Care Unit. JAMA. 2017 Jan 17;317(3):290-300. doi: 10.1001/jama.2016.20328. PMID 28114553